CLINICAL TRIAL: NCT04653467
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG4399 in Adult, Healthy, Male Subjects
Brief Title: A Study to Evaluate How Well Single and Multiple Doses of GLPG4399 Are Tolerated in Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG4399-CL-101
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part 1: a randomized, double-blind, single ascending dose (SAD), Part 2: a randomized, double-blind, multiple ascending dose (MAD) escalation and Part 3 and 4: an open-label, randomized, crossover rBA and food-effect (FE) part.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GLPG4399 SAD (Experimental): Single doses of GLPG4399 at up to 6 dose levels in ascending order
  Interventions: Drug: GLPG4399 oral suspension
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo
- GLPG4399 MAD (Experimental): Multiple ascending doses of GLPG4399
  Interventions: Drug: GLPG4399 oral suspension
- Placebo MAD (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo
- GLPG4399 FE-rBA (Experimental): Single dose of GLPG4399 in fed and fasted state
  Interventions: Drug: GLPG4399 oral suspension; Drug: GLPG4399 capsules
- GLPG4399 FE (Experimental): Single dose of GLPG4399 in fed and fasted state
  Interventions: Drug: GLPG4399 oral suspension

INTERVENTIONS:
Drug: GLPG4399 oral suspension — GLPG4399 for oral administration
  Arms: GLPG4399 FE; GLPG4399 FE-rBA; GLPG4399 MAD; GLPG4399 SAD
Drug: GLPG4399 capsules — GLPG4399 for oral administration
  Arms: GLPG4399 FE-rBA
Drug: Placebo — Placebo oral suspension
  Arms: Placebo MAD; Placebo SAD

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single (part 1) and multiple ascending (part 2) oral doses of GLPG4399, in adult, healthy, male subjects. In addition, the effect of food and the relative bioavailability (rBA) of GLPG4399, will be evaluated (part 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests, available at screening and prior to randomization. Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be no greater than 1.5x upper limit of normal range (ULN). Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.
* Subject must be able and willing to comply with restrictions on prior and concomitant medication
* Negative screen for drugs (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants) and alcohol.
* Able and willing to comply with the clinical study protocol (CSP) requirements and to sign and date the ICF as approved by the Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to any screening evaluations.

Exclusion Criteria:

* Subject has a history of any drug allergies.
* Known hypersensitivity to investigational product (IP) ingredients or history of a significant allergic reaction to IP ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IP.
* Subject testing positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as detected by real-time polymerase chain reaction (RT-PCR) or subjects who have been in contact with SARS-CoV-2 infected individuals in the 2 weeks prior to first dosing of IP. Subjects presenting any signs or symptoms of SARS-CoV-2 infection as detected at screening and/or baseline following careful physical examination (e.g. cough, fever, headaches, fatigue, dyspnea, myalgia, anosmia, dysgeusia, anorexia, sore throat, etc.) will also be excluded. In addition, any other locally applicable standard diagnostic criteria may also apply to diagnose SARS-CoV-2 infection.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus (HIV) infection).
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first dosing of the IP.
* Presence or sequelae of gastrointestinal, liver, kidney (estimated glomerular filtration rate (eGFR) <=90 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within the past 5 years prior to screening with the exception of excised and curatively treated non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin which is considered cured with minimal risk of recurrence.
* Vital sign abnormalities (systolic blood pressure <90 or >140 mmHg, diastolic blood pressure <60 or >90 mmHg, or heart rate <60 or >100 bpm) at screening.
* History or presence of clinically significant abnormalities detected on 12-lead ECG of either rhythm or conduction e.g. known long QT syndrome or a QT interval corrected for heart rate using Fridericia's formula: QTcF = QT/RR1/3 (QTcF) >450 ms detected on the 12-lead ECG. A first-degree atrioventricular block will not be considered as a significant abnormality.
* Personal or family history of long QT syndrome or unexplained sudden cardiac death in a first-degree relative.
* Male subjects with female partners of child bearing potential not willing to comply with the contraceptive methods
* Significant blood loss (including blood donation [>450 mL]), or transfusion of any blood product within 12 weeks prior to (first) dosing.
* Treatment with any drug known to have a potential for major organ toxicity in the last 3 months before first dosing of the IP.
* Treatment with any medication (including over-the-counter (OTC) and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing of IP.
* Active drug abuse or alcohol abuse (alcohol abuse defined as regular weekly intake of more than 14 units1) within 2 years prior to first IP administration.
* Active smoker and/or has used e-cigarettes, nicotine, or nicotine-containing products within the past 6 months before the first IP administration.
* Regular consumption of a large quantity of caffeinated coffee, tea (>6 cups per day) or equivalent.
* Concurrent participation or participation in a drug, drug/device or biologic investigational research study within 12 weeks or 5 half-lives of the IP, whichever is longer, prior to first dosing.
* Investigator or other study staff or relative thereof who is directly involved in the conduct of the study.
* Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From screening through study completion, an average of 6 months
  To evaluate the safety and tolerability of single and multiple ascending oral doses of GLPG4399 in adult, healthy, male subjects.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG4399 | Between Day 1 pre-dose and Day 33
  To evaluate the pharmacokinetics (PK) of single and multiple ascending oral doses of GLPG4399, in adult, healthy, male subjects.
Area under curve (AUC) of GLPG4399 | Between Day 1 pre-dose and Day 33
  To evaluate the pharmacokinetics (PK) of single and multiple ascending oral doses of GLPG4399, in adult, healthy, male subjects.
Terminal elimination half-life (t1/2) of GLPG4399 | Between Day 1 pre-dose and Day 33
  To evaluate the pharmacokinetics (PK) of single and multiple ascending oral doses of GLPG4399, in adult, healthy, male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- Altasciences Montreal, Mount Royal, Canada

IPD SHARING:
Plan to Share IPD: No